CLINICAL TRIAL: NCT01714232
Title: Evaluation of Blood Glucose Meter Systems - Contour® PLUS Study
Brief Title: Evaluation of Blood Glucose Meter Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2012-008-01
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Results first posted 2013-12-27 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Staff Test BGMSs (Experimental): All testing and lancing were performed by the study staff; subjects did not perform any lancing or self-testing in this study. Study Staff lanced the fingers of subjects and tested the blood samples using five Blood Glucose Monitoring Systems (BGMS): Contour® PLUS BGMS; OneTouch® SelectSimple™ BGMS; Accu-Chek® Performa BGMS; Accu-Chek® Active BGMS; Freestyle Freedom® BGMS.
  Interventions: Device: Contour® PLUS BGMS; Device: OneTouch® SelectSimple™ BGMS; Device: Accu-Chek® Performa BGMS; Device: Accu-Chek® Active BGMS; Device: Freestyle Freedom® BGMS

INTERVENTIONS:
Device: Contour® PLUS BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: OneTouch® SelectSimple™ BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Accu-Chek® Performa BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Accu-Chek® Active BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Freestyle Freedom® BGMS — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes and without diabetes (up to 10% of subjects without diabetes were included). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).

SUMMARY:
The purpose of this study was to evaluate the performance of a Bayer Blood Glucose Monitoring System (BGMS) and four additional Blood Glucose Monitoring Systems (BGMS) from other manufacturers. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the performance of a Bayer Blood Glucose Monitoring System (BGMS) and four additional Blood Glucose Monitoring Systems (BGMS) from other manufacturers. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer). Performance of the five systems were evaluated across the glucose range of the BGMSs using capillary blood. All testing and lancing were performed by study staff and some samples were tested from subject fingertips. Additionally, some blood samples were glycolyzed to lower the glucose concentration levels and glucose solution was added to other samples to raise glucose concentration levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age or older
* Willing to complete all study procedures

Exclusion Criteria:

* Blood Borne infections like hepatitis or HIV or infections such as tuberculosis
* Hemophilia or any other bleeding disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Simmons, MD, Principal Investigator — Ascensia Diabetes Care
Locations (1):
- Bayer HealthCare LLC, Diabetes Care, Mishawaka, Indiana, United States

REFERENCES:
- [Derived] Pardo S, Dunne N, Simmons DA. A comparison of bolus insulin dose errors based on results of a clinical trial of five blood glucose monitoring systems. Ther Deliv. 2019 Dec;10(12):793-799. doi: 10.4155/tde-2019-0047. Epub 2019 Dec 2. PMID 31789119
- [Derived] Dunne N, Viggiani MT, Pardo S, Robinson C, Parkes JL. Accuracy Evaluation of CONTOUR((R))PLUS Compared With Four Blood Glucose Monitoring Systems. Diabetes Ther. 2015 Sep;6(3):377-88. doi: 10.1007/s13300-015-0121-3. Epub 2015 Jul 14. PMID 26169192

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Staff Test BGMSs: All testing and lancing were performed by the study staff; subjects did not perform any lancing or self-testing. Study Staff lanced the fingers of subjects and tested the blood samples using five Blood Glucose Monitoring Systems (BGMS): Contour® PLUS BGMS; OneTouch® SelectSimple™ BGMS; Accu-Chek® Performa BGMS; Accu-Chek® Active BGMS; Freestyle Freedom® BGMS.
Period: Overall Study
Arm/Group | Study Staff Test BGMSs
Started | 106
Completed | 106
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 106
Age, Customized [Median (Full Range); unit: years] | 60 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 106

OUTCOME MEASURES:

1. Primary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) Across the Overall Tested Glucose Range
Description: Using the overall Blood Glucose (BG) range (27 to 460 mg/dL), the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI laboratory reference values were compared. MARD was calculated from the sum of all |(BG meter)-(BG reference)|/(BG reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all 5 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD values indicate smaller differences between meter value and the reference value. Higher MARD values indicate higher differences between meter value and the reference value.
Time Frame: 8 hours
Population: 314 BG results possible for each BGMS (318-4=314). Staff collected 3 capillary samples from each subject-total 318 samples. One subject hematocrit(56%) was above the study evaluable limit 55%, so that subject's 3 samples were not analyzed. One sample from another subject was below meter operating limit (12.3mg/dL) so it was not analyzed.
Measure: Mean (Standard Error); unit: Percent Difference
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 105
Percent Difference
  Contour® PLUS BGMS | 3.3 (0.31)
  Accu-Chek® Performa BGMS | 4.9 (0.31)
  Accu-Chek® Active BGMS | 5.8 (0.31)
  OneTouch® SelectSimple™ BGMS | 10.7 (0.31)
  Freestyle Freedom® BGMS | 15.3 (0.31)

2. Secondary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) in the Low Glucose Range(<=80 mg/dL)
Description: Using fresh and glycolyzed samples with Blood Glucose (BG) <=80 mg/dL, the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI laboratory reference values were compared. MARD was calculated from the sum of all |(BG meter)-(BG reference)|/(BG reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all 5 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD values indicate smaller differences between meter value and the reference value. Higher MARD values indicate higher differences between meter value and the reference value.
Time Frame: 8 hours
Population: Same number (93) of BG results was possible for each BGMS. Staff collected 3 capillary samples from each subject (total 314), of which 93 samples were less than or equal to 80 mg/dL.
Measure: Mean (Standard Error); unit: Percent Difference
Units Other Than Participants: BG Test Results
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 105
Number analyzed (BG Test Results) | 93
Percent Difference
  Contour® PLUS BGMS | 3.4 (0.60)
  Accu-Chek® Performa BGMS | 4.2 (0.60)
  Accu-Chek® Active BGMS | 6.4 (0.60)
  OneTouch® SelectSimple™ BGMS | 13.3 (0.60)
  Freestyle Freedom® BGMS | 17.7 (0.60)

3. Secondary Outcome: MARD (Mean Absolute Relative Difference Between BGMS Results and Reference Method Results) in the High Glucose Range (>180 mg/dL)
Description: Using samples with Blood Glucose >180 mg/dL, the Mean Absolute Relative Differences (MARD) between the BGM System readings and the YSI laboratory reference values were compared. MARD was calculated from the sum of all |(BG meter)-(BG reference)|/(BG reference) assessments, divided by the number of assessments, then multiplied by 100(%). Each evaluable sample was tested on all 5 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MARD values indicate smaller differences between meter value and the reference value. Higher MARD values indicate higher differences between meter value and the reference value.
Time Frame: 8 hours
Population: Same number (113) of BG results was possible for each BGMS. Staff collected capillary samples from each subject as described in primary objective population description, of which 113 samples were greater than 180 mg/dL.
Measure: Mean (Standard Error); unit: Percent Difference
Units Other Than Participants: BG Test Results
Arm/Group | Study Staff Test BGMSs
Number analyzed (Participants) | 105
Number analyzed (BG Test Results) | 113
Percent Difference
  Contour® PLUS BGMS | 3.3 (0.50)
  Accu-Chek® Performa BGMS | 5.9 (0.50)
  Accu-Chek® Active BGMS | 5.7 (0.50)
  OneTouch® SelectSimple™ BGMS | 9.8 (0.50)
  Freestyle Freedom® BGMS | 14.1 (0.50)

ADVERSE EVENTS:
Arm/Group | Study Staff Test BGMSs
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 3/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Staff Test BGMSs (N=106)
Hypoglycemia (Endocrine disorders) | 3 (3) — Adverse events were mild, anticipated, non-device related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes